CLINICAL TRIAL: NCT06011434
Title: Testing a Conversation Aid on Mammography Screening for Clinicians and Women 75 and Older in Practice
Brief Title: Testing Conversation Aid in Practice
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mara Schonberg, Principal Investigator, Beth Israel Deaconess Medical Center
Other Study IDs: 23-201; R01AG065311 (NIH)
Record Dates: First submitted 2023-08-08; First posted 2023-08-25 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Mammography; Breast Cancer Screening; Mammography Screening
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patient: Conversation Aid On Mammography Screening: Participants will complete study procedures as follows:
  * Pretest questionnaires.
  * PCP Appointment with introduction to conversation aid website.
  * Post-test questionnaires within two weeks of PCP visit.
  Interventions: Behavioral: Mammography Screening Conversation Aid
- Family: Conversation Aid On Mammography Screening: Caretakers/Family members to participants will complete study procedures as follows:
  * Pretest questionnaires.
  * Attend with participant PCP Appointment with introduction to conversation aid website.
  * Post-test questionnaires within two weeks of PCP visit.
  Interventions: Behavioral: Mammography Screening Conversation Aid
- Clinician: Conversation Aid On Mammography Screening: Clinicians will complete study procedures as follows:
  * Pretest questionnaires.
  * Post-test questionnaires.
  Interventions: Behavioral: Mammography Screening Conversation Aid

INTERVENTIONS:
Behavioral: Mammography Screening Conversation Aid — Web-based, "Decide Together" conversation aid designed to be used by PCP and participant for shared decision making and to provide information on the benefits and harms of mammography screening as well as educational talking points.

SUMMARY:
The goal of this research study is to develop and test a website to help primary care providers (PCPs) discuss the pros and cons of mammography with women aged 75 and older and to help participants make decisions about mammography.

DETAILED DESCRIPTION:
This research study is to conduct a pilot pretest-posttest trial to learn if providing a web-based conversation aid (CA) on mammography screening to 36 primary care providers facilitates shared decision making (SDM) and 8 medical assistants with 190 of their patients (2-3 per PCP) aged 75-89 years and 23 involved family members.

Research procedures include screening for eligibility, questionnaires, and clinic visits.

Participation in this research study is expected to last about 4 months.

It is expected about 90 participants, 23 participant family members, 36 primary care providers, and 8 medical assistants will participant in this research study.

The National Institute on Aging is supporting this research study by providing funding.

ELIGIBILITY:
Participant Inclusion Criteria:

* English-speaking
* Aged 75 - 89 years
* Seen by an attending-level (non-resident) seen at the recruitment practices who have the -Ability and willingness to provide verbal consent.

Participant Family Members Inclusion Criteria:

* Family member of patient that has agreed to participate in the study
* Age >18
* English speaking
* Ability and willingness to provide verbal consent

Primary Care Provider Inclusion Criteria:

* Non-resident physician, nurse practitioner, or physician assistant

  ->18 years old
* English speaking
* Cares for a panel of patients that includes women >75 years at one of the recruitment practices
* Ability and willingness to provide verbal consent

Participant Exclusion Criteria:

* Last mammogram <6 or >30 months (so that participants may be contemplative of their next mammogram)
* History of dementia
* Incapacity for informed consent
* History of invasive or non-invasive breast cancer
* Last mammogram was abnormal
* Non-English speaking
* Already chose to stop being screened (documented in medical records or scores of 1-3 [do not intend to be screened] on a validate 15 point intentions to be screened scale.)
* PCP unwilling to have patient participate
* In hospice
* PCP not willing to participate
* Psychiatric illness situations that would limit compliance with study requirements

Participant Family Member Exclusion Criteria:

* Age <18
* Non-English speaking
* Psychiatric illness situations that would limit compliance with study requirements

Primary Care Provider Exclusion Criteria:

* Resident physician
* Psychiatric illness situations that would limit compliance with study requirements

Ages: 75 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Study Population: Primary care practices at Beth Israel Deaconess Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 157 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Intentions For Screening Questionnaire | 1-12 weeks for pretest and 1 - 4 weeks for posttest, up to 4 months.
  Assessed by the Intentions for Screening questionnaire, a 15-point validated measure (1 to 15) to assess one's leaning towards an option with scores of 1=no, 8= unsure, and 15=yes.

SECONDARY OUTCOMES:
Shared Decision Making (SDM) Questionnaire | 1-12 weeks for pretest and 1 - 4 weeks for posttest, up to 4 months.
  Assessed by the validated, 9-item SDM questionnaire. Each item will be scored on a 6-point Likert scale with answers ranging from 0 "completely disagree" to 6 "completely agree." A total score will range from 9 - 54.
Decisional Conflict Questionnaire | 1-12 weeks for pretest and 1 - 4 weeks for posttest, up to 4 months.
  Assessed by the Decisional Conflict Questionnaire, a validated, 16 item scale scored on a 5-point Likert scale. Answers range from 1 "Strongly Agree" to 0 "Neutral" to 4 " Strongly Agree" with each score ranging from 0 - 4 points. A total is calculated by [sum of scores/16] x 25=scale 0-100).
Role In Decision (Decision Making Preferences Questionnaire) | 1-12 weeks for pretest and 1 - 4 weeks for posttest, up to 4 months.
  Controlled preferences scale Assessed by the Decision Making Preferences questionnaire which includes 5 response categories (see comments). We will group the 5-items into 3 categories (patient prefers to make the decision, patient prefers the PCP makes the final decision, the patient prefers to share the decision with the PCP). This scale is commonly used to assess a participant's preferred involvement in decision making.
Participant Knowledge Questionnaire | 1-12 weeks for pretest and 1 - 4 weeks for posttest, up to 4 months.
  Assessed by the participant knowledge questionnaire, comprised of 10 True/False questions. Total score will be reported as a mean percentage of the number of questions answered correctly.
Mammogram Attitudes Questionnaire | 1-12 weeks for pretest and 1 - 4 weeks for posttest, up to 4 months.
  Assessed by the mammogram attitudes questionnaire, comprised of 3 questions graded on a 7-point Likert scale with answers ranging from 1 "Completely Unnecessary/Harmful/Unpleasant" to 7 "Completely Necessary/Beneficial/Pleasant. Scores will be summed and a total score will range from 3 - 21.
Mammogram Perceived Norms Questionnaire | 1-12 weeks for pretest and 1 - 4 weeks for posttest, up to 4 months.
  Assessed by the mammogram norms questionnaire, comprised of 2 questions graded on a 7-point Likert scale with answers ranging from 1 "Strongly Disagree" to 7 "Strongly Agree." Scores will be summed and a total score will range from 2 - 14.
Clinician Self-Efficacy Scale | 1-12 weeks for pretest and 1 - 4 weeks for posttest, up to 18 months.
  Assessed by the clinician self-efficacy subscale of the Shared Decision Making (SDM) Questionnaire, which measures clinician self-efficacy to engage older women in shared decision making around mammography screening and is comprised of 5 questions graded on a 7-point Likert scale with answers ranging from 1 "Strongly Disagree/Easy" to 7 "Strongly Agree/Difficult." A total score will range from 5 to 35.
Clinician Attitudes Scale | 1-12 weeks for pretest and 1 - 4 weeks for posttest, up to 18 months.
  Assessed by the clinician attitudes Subscale of the Share Decision Making (SDM Questionnaire which is comprised of 4 questions about clinician attitudes towards mammography screening and graded on a 7-point Likert scale with scores ranging from "1 "Unnecessary/Harmful/Unpleasant/Worthless" to 7 "Necessary/Beneficial/Pleasant/Useful." A total score will range from 4 - 28.
Clinician Perceived Norms Scale | 1-12 weeks for pretest and 1 - 4 weeks for posttest, up to 18 months.
  Assessed by the clinician perceived norms subscale of the Shared Decision Making (SDM) Questionnaire which is comprised of 4 questions about clinician perceived norms around mammography screening and graded on a 7-point Likert scale with answers ranging from 1 "Strongly Disagree" to 7 "Strongly Agree." A total score will range from 4 - 28.

CONTACTS AND LOCATIONS:
Overall Officials: Mara Schonberg, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu